CLINICAL TRIAL: NCT00160485
Title: Glyburide Compared to Insulin in the Management of White's Classification A2 Gestational Diabetes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Active Duty principle investigator currently deployed
Sponsor: Tripler Army Medical Center (U.S. Federal Agency)
Responsible Party: COL Elizabeth Golladay Spooner, MD, Tripler Army Medial Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAMC 16H04
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2011-07

CONDITIONS: Gestational Diabetes
Keywords: Gestational Diabetes; Pregnancy; Glyburide; Insulin
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance | interventions — Glyburide; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Glyburide,gestational diabetes, maternal complications, neonatal complications
  Interventions: Drug: Glyburide
- 2 (Active Comparator): Insulin, gestational diabetes, maternal complications, neonatal outcomes
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Glyburide — dosage required to obtain adequate glucose control
  Arms: 1
Drug: Insulin — variable dosage to obtain glucose control
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the oral administration of glyburide is as effective as insulin in the treatment of gestational diabetes.

1. SYNOPSIS: Infants born to mothers with gestational diabetes(GDM) are at risk for a variety of adverse perinatal outcomes including macrosomia with subsequent birth trauma and cesarean delivery, neonatal hypoglycemia, polycythemia, jaundice, hypocalcemia, respiratory depression and newborn intensive care unit admission. These adverse outcomes are thought to be related to the degree of maternal hyperglycemia during pregnancy. Women with GDM are typically treated with insulin to lower blood glucose levels to as near-normal as possible. A single randomized trial has suggested that the oral sulfonylurea, glyburide is a clinically effective and safe alternative to insulin therapy.
2. Many obstetric care providers have adopted the use of glyburide in the routine management of gestational diabetes. The American College of Obstetrics and Gynecology and the American Diabetic Association both state that further studies are needed in a larger patient population before the use of newer oral hypoglycemic agents can be supported for use in pregnancy.
3. STATUS: Previous studies have demonstrated that there is no maternal-fetal transfer of glyburide and when compared to insulin is an effective alternative to insulin. Additionally, a published cost analysis concluded that glyburide is significantly less costly than insulin for the treatment of GDM. The benefits of an oral agent for the management of gestational diabetes include less discomfort for the patient in drug administration, lower requirement for patient education in the administration of injectable medications and less chance of error in dosing. Our study population is more ethnically diverse and our incidence of large for gestational age infants is lower than in the largely Hispanic population studied by Langer et al. Many obstetricians, including ourselves, apply different criteria than Langer for diagnosing gestational diabetes , and for deciding when to institute insulin therapy. It is our goal to confirm the prior single study concerning the safety and efficacy of glyburide in reducing the complications of GDM utilizing a more ethnically diverse population with more realistic goals in glycemic control. To this end we will add to the medical literature supporting this alternative therapy to insulin.

DETAILED DESCRIPTION:
PLAN: Women who present for prenatal care are routinely screened for gestational diabetes (GDM) with a one-hour 50gm oral glucose challenge test (GCT). This screening occurs at the first prenatal visit if risk factors (marked obesity, prior pregnancy affected by GDM, prior macrosomic infant, glycosuria, strong family history of diabetes) for GDM are identified on intake history. If no risk factors for GDM are identified or if initial screening is negative, the GCT is administered between 24-28 weeks gestation. At our institution, the GCT is considered positive if, one hour after ingestion of a 50gm oral glucose solution, the serum glucose is greater than or equal to 135mg/dl. This screening cutoff varies among medical treatment facilities. Positive screening tests are followed by a diagnostic oral glucose tolerance test (GTT). A positive diagnosis requires that two or more thresholds be met or exceeded. Women with the diagnosis of gestational diabetes will receive dietary counseling and instruction on the performing capillary glucose from a by a nurse educator. If > 20% of recorded home glucose values are in excess of target range following initiation of appropriate diet, women will be offered enrollment into the study.

All women who agree to participate in the study will have an ultrasound performed to confirm gestational age and rule out fetal anomalies, a serum glycosylated hemoglobin A1C to assist in excluding preexisting diabetes and a fasting insulin level to assist in determining degree of insulin resistance. A serum glycosylated hemoglobin A1C will be repeated upon admission for delivery. Subjects randomized into standard therapy insulin arm will have their insulin dose calculated by established standards. Dosing is based upon a 2 shot combined dose with long acting and short acting insulin given prior to breakfast and dinner. If the fasting glucose values remain elevated the dinner NPH will be moved to bedtime. Subcutaneous administration is recommended in a consistent anatomic region, preferably the abdomen.

Insulin will be adjusted on a weekly basis in order to maintain optimal glucose control. Women assigned to receive glyburide will begin with 2.5mg orally with the morning meal. Glyburide dosage will be increased weekly as indicated to a maximum daily dose of 20mg to achieve glucose control. If the patient continues to have elevated fasting glucose the may be split to 12 hr intervals. If maximum daily dose of glyburide does not result in reaching the threshold values, patients will be administered insulin however data will be analyzed on an intent-to-treat basis.

Upon admission for delivery additional maternal blood will be collected for hemoglobin A1C, and glyburide levels. These values will be utilized to determine efficacy of treatment and for comparison to fetal umbilical cord values.

At delivery fetal blood from the umbilical cord will be collected for glucose, hematocrit, insulin level and, in a representative sample, glyburide level. These values will be utilized to determine whether insulin or glyburide provides superior efficacy in maintaining these values within normal limits. Cord blood glyburide levels will be obtained in a representative sample of exposed subjects.

When clinically indicated labs are performed by the pediatrician on the newborn, such as heel stick glucose for hypoglycemia, bilirubin levels for neonatal jaundice, calcium levels for suspected hypocalcemia, these values will be obtained by review of the newborn record.

In all gestational diabetics, post partum assessment of diabetic status will be assessed with either a fasting glucose determination or a 2hr glucose tolerance test .

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over age 18 who fail to achieve adequate glucose control on diet therapy alone.

Exclusion Criteria:

* Delivery planned at other than a participating medical treatment facility.
* Women with preexisting diabetes mellitus or diabetic ketoacidosis.
* Hypersensitivity to study medications
* Underlying vascular disease or medical condition known to affect fetal growth or drug clearance such as: severe chronic hypertension, systemic lupus erythematosis, chronic renal insufficiency, hepatic disease, antiphospholipid antibody syndrome or thrombophilia.
* Fetal anomalies identified on ultrasound prior to initiation of therapy.
* Fetal aneuploidy.
* Diagnosis of GDM made after 32 weeks gestation (fetal growth pattern may be impossible to affect after this gestational age.)
* Use of supplemental herbal/nutraceuticals containing chromium, garlic, gymnema (may cause hypoglycemia).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-06; Primary Completion 2009-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Newborn birth weight | mid study

SECONDARY OUTCOMES:
Gestational age at delivery | Completion of study
Method of delivery (cesarean, forceps, vacuum, spontaneous) | completion of study
Complications of delivery (shoulder dystocia, birth injury, 4th degree vaginal laceration) | completion of study
Newborn intensive care unit admission | mid study
Congenital anomalies of the newborn | completion of study
Incidence of neonatal metabolic derangement | completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth G Spooner, MD, Principal Investigator — Tripler Army Medical Center
Locations (1):
- Tripler Army Medical Center, Honolulu, Hawaii, United States